CLINICAL TRIAL: NCT07181291
Title: Pulsed Field or Cryoballoon Pulmonary Vein Isolation for Atrial Fibrillation in Heart Failure (a Propensity Score Matched Comparison)
Brief Title: Pulsed Field or Cryoballoon Pulmonary Vein Isolation for Atrial Fibrillation in Heart Failure
Status: Active, not recruiting | Type: Observational
Sponsor: St. Josefs-Hospital Wiesbaden GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: PFA vs CRYO for AF-HFrEF
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cryoballoon pulmonary-vein isolation: Electrical isolation of the pulmonary-veins using cryoenergy
  Interventions: Procedure: PVI
- Pulsed field pulmonary-vein isolation: Electrical isolation of the pulmonary-veins using pulsed field energy
  Interventions: Procedure: PVI

INTERVENTIONS:
Procedure: PVI — pulmonary-vein isolation

SUMMARY:
Patients with atrial fibrillation (AF) and heart failure with reduced left ventricular ejection fraction (HFrEF) are at particularly high cardiovascular risk. Rhythm-control by means of catheter-based pulmonary vein isolation (PVI) reduces all-cause mortality and rehospitalization for worsening heart failure in these patients. Considering the globally increasing use of the novel "pulsed-field ablation", it is necessary to determine whether this technique can be performed with the same safety and efficacy as the established cryoballoon ablation (CBA) in this critically ill patient population.

This research project aims to retrospectively compare, in a multicenter study, PVI using PFA and CBA in patients with AF and concomitant HFrEF based on pre-collected pseudonymized patient data through propensity score matching.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with paroxysmal or persistent AF and echocardiographically confirmed HFrEF (LVEF ≤ 40%)
2. Patients who underwent their first PVI using pulsed field or cryoballoon ablation as part of clinical routine
3. Patients with regular follow-up via 12-lead ECG or Holter ECG following PVI
4. Patients with at least three months of follow-up

Exclusion Criteria:

1. Patients who did not undergo pulsed field or cryoballoon ablation for first-time PVI
2. Patients with LVEF > 40%
3. Patients who declined the use of their data during initial collection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation and heart failure (LVEF ≤ 40%)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a clinical recurrence of any atrial arrhythmia (AF, atrial flutter, atrial tachycardia) occurring more than 8 weeks post-intervention | 12 months
  First documented clinical recurrence of any atrial arrhythmia

SECONDARY OUTCOMES:
Number of patients with a rehospitalization (≥ 1 night) due to atrial arrhythmia/ re-ablation or electrical cardioversion starting from day 1 post index procedure | 12 months
Number of patients with a rehospitalization (≥ 1 night) due to worsening heart failure | 12 months
Death from any cause | 12 months
Number of subjects with procedure-associated complications | 30 days
  Death, Major bleeding (criteria per Bleeding Academic Research Consortium ≥2, treatment-requiring groin complications (including AV fistula, aneurysm, or dissection), pericardial effusion/tamponade, non-fatal stroke/transient ischemic, attack, temporary or persistent phrenic nerve palsy, homeless

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Ehrlich, MD, Principal Investigator — St. Josefs-Hospital Wiesbaden GmbH
Locations (10):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Montreal Heart Institute, Montreal, Quebec
- Germany (7):
  - Vivantes Klinikum am Urban, Berlin
  - Universitätsklinikum Frankfurt am Main, Frankfurt am Main
  - Klinikum Fürth, Fürth
  - Evangelisches Krankenhaus Hagen-Haspe, Hagen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - St. Josefs-Hospital Wiesbaden, Wiesbaden
- Maastricht University Medical Center Plus, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No